CLINICAL TRIAL: NCT03308747
Title: Effects of Low-grade Systemic Inflammation on Muscle Protein Synthesis and Breakdown in the Aged Skeletal Muscle.
Brief Title: Inflammaging and Muscle Protein Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Associate Professor, University of Thessaly
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: INFLAMMAGING-UTH
Record Dates: First submitted 2017-10-02; First posted 2017-10-13 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2017-10

CONDITIONS: Inflammaging; Sarcopenia
Keywords: Low-grade systemic inflammation; Muscle protein synthesis; Proteasome activation; Anabolic signaling; Aging; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High systemic inflammation (Experimental): Individuals assigned in the high systemic inflammation group will be characterized by IL6: ≥ 1.7 pg/ml and hs-CRP: > 2.0 mg/L.
  Interventions: Dietary Supplement: Instantized Whey Protein Isolate
- Low systemic inflammation (Active Comparator): Individuals assigned in the high systemic inflammation group will be characterized by IL6: < 1.7 pg/ml and hs-CRP: < 1.0 mg/L.
  Interventions: Dietary Supplement: Instantized Whey Protein Isolate

INTERVENTIONS:
Dietary Supplement: Instantized Whey Protein Isolate — 0,4 g of whey protein isolate/kg body weight will be ingested as a bolus of 250 ml immediately after the resistance exercise bout.

SUMMARY:
The development of a low-grade, chronic, systemic inflammation observed in the elderly (inflammaing) has been associated with increased risk for skeletal muscle wasting, strength loss and functional impairments. According to studies performed in animals and cell cultures increased concentrations of pro-inflammatory cytokines such as IL-6 and TNF-α as well as increased levels of hs-CRP lead to elevated protein degradation through proteasome activation and reduced muscle protein synthesis (MPS) via downregulation of the Akt-mTOR signaling pathway. However, evidence regarding the effects of inflammaging on skeletal muscle mass in humans is lacking. Thus, the present study will compare proteasome activation and the protein synthetic response in the fasted and postprandial period between older adults with increased systemic inflammation and their healthy control counterparts.

DETAILED DESCRIPTION:
A total number of > 60 male, older adults aged 63-73 years will be initially screened for systemic levels of hs-CRP and IL-6. Of these, 24 individuals that will comply with the study criteria will be allocated to either a High (IL6: ≥ 1.7 pg/ml; hs-CRP: > 1.0 mg/L) (n=12) or a Low (IL6: < 1.7 pg/ml; hs-CRP: < 1.0 mg/L) (n=12) systemic inflammation group. Approximately 2 weeks before the experimental trial, anthropometry, resting metabolic rate (RMR), body composition (with DXA), sarcopenia status, functional capacity and the knee-extension one repetition maximum (1RM) will be assessed in individuals from both groups. In addition, levels of habitual physical activity will be assessed using accelerometry (over a 7-day period) and daily dietary intake will be monitored through 7-day diet recalls in all participants. 1 week before the experimental day an oral glucose tolerance test (OGTT) will be also performed over a 2-hour period, with blood sampling every 15min during the first hour and every 30min during the second hour. The day before the experimental trial, participants will consume 150ml of D2O 70% atom as a bolus. In the experimental day, participants will arrive at the laboratory after an overnight fast and a baseline blood sample and a muscle biopsy from vastus lateralis muscle will be collected. Immediately after, participants will perform 8 sets with 10 repetitions at 80% of 1RM and 2 min rest between each set, on a knee-extension machine. After exercise, they will ingest 0.4 g whey protein isolate/kg body weight as single bolus and then they will remain in a sitting position over a 3-hour period. Blood samples will be collected every 30min during the 3-hour postprandial period while a second muscle biopsy will be obtained at 3h.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers.
* BMI ≥18.5 & BMI ≤ 35 kg/m2.
* Moderately active but with no regular participation in heavy resistance exercise within the last 6 months.
* Absence of chronic disease (i.e. cancer, metabolic, cardiac, or neurological diseases).
* Free and independently living.

Exclusion Criteria:

* Organ failure (unstable, renal, respiratory, liver).
* Chronic use of corticosteroid medication.
* Recent use of antibiotics.
* Presence of frailty.
* Body weight variation over the past 6mo > 10% or weight loss of more than 3kg in the last 3 months.
* Use of anti-inflammatory or lipid-lowering medication (i.e., statins).
* Use of medication interacting with muscle metabolism.

Ages: 63 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Systemic inflammation | At baseline.
  Levels of systemic inflammation will be assessed by measuring serum levels of hs-CRP, IL-6 and TNF-α.
Change in muscle protein synthesis (MPS) | At baseline and 180 min following protein ingestion.
  Using deuterium oxide (D2O) 70% atom administration. Individuals will consume a single bolus of 150ml D20 the day before the clinical trial and muscle biopsy samples, collected before and after the exercise bout and protein ingestion, will be analyzed for isotopic measurement using GC-P-IRMS.
Change in intracellular signaling proteins in muscle | At baseline and 180 min following protein ingestion.
  Phosphorylation levels of Akt, mammalian target of rapamycin (mTOR), p70S6K and ribosomal protein S6 (rpS6) will be measure using western blotting.
Change in proteasome activities in muscle | At baseline and 180 min following protein ingestion.
  Chymotrypsin-like (CT-L), caspase-like (C-L) and trypsin-like (T-L) proteasome activities will be assayed with hydrolysis of the fluorogenic peptide LLVY-AMC, LLE-AMC and LSTR-AMC, respectively.
Change in protein expression level of proteasome subunits | At baseline and 180 min following protein ingestion.
  Immunoblot analysis will be used to detect protein expression levels of proteasome (β5, β2 and β1) and immunoproteasome (β5i, β2i and β1i) subunits.

SECONDARY OUTCOMES:
Resting metabolic rate (RMR) | At baseline.
  RMR will be assessed after an overnight fast with participants in a supine position following a 15-min stabilization period by taking 30 consecutive 1-min VO2/CO2 measurements using a portable open-circuit indirect calorimeter with a ventilated hood system following a standard calibration protocol.
Physical activity | Over a 7-day period at baseline.
  Level of habitual physical activity will be assessed using accelerometry (ActiGraph GT3X-BT accelerometer).
Dietary intake | Over a 7-day period at baseline.
  Daily dietary intake will be assessed using 7-day diet recalls.
Reduced glutathione in blood | At baseline.
  Concentration of reduced glutathione will be measured in red blood cells
Oxidized glutathione in blood | At baseline.
  Concentration of oxidized glutathione will be measured in red blood cells
Protein carbonyls in serum | At baseline.
  Concentration of protein carbonyls will be measured in serum.
Total antioxidant capacity | At baseline.
  Total antioxidant capacity will be measured in serum
Malondialdehyde in serum | At baseline.
  Concentration of malondialdehyde will be measured in serum.
White blood cell count in blood | At baseline.
  White blood cell count will be measured in blood.
Insulin sensitivity | At baseline.
  Insulin sensitivity will be assessed through an oral glucose tolerance test (OGTT) which involve ingesting glucose solution (75 g) with 5ml arterialized venous blood samples drawn at baseline and every 15 min during the first hour and every 30 min during the second hour over a 2-hour period.
Glucose concentration in blood | At baseline and at 30 min, 60 min, 90 min, 120 min, 150 min and 180 min following protein ingestion.
  Glucose concentration will be measured in plasma during the clinical trial.
Insulin concentration in blood | At baseline and at 30 min, 60 min, 90 min, 120 min, 150 min and 180 min following protein ingestion.
  Insulin concentration will be measured in plasma during the clinical trial.
Body composition | At baseline
  Body composition will be measured using a dual-energy x-ray absorptiometry scanner (DEXA).
Body Mass Index (BMI) | At baseline
  Calculated as body mass (kg) divided by the height (m) squared.
Skeletal muscle index | At baseline
  Calculated as an appendicular lean mass (kg) divided by height (m) squared.
Grip strength | At baseline
  Using handgrip dynamometry (left and right arm) in a sitting position.
Functional performance | At baseline
  Functional performance will be assessed using the Short Physical Performance Battery (SPPB).
Lower limb muscle strength | At baseline
  Will be assessed by defining the 1 repetition maximum (1RM) on a knee-extension machine.

CONTACTS AND LOCATIONS:
Overall Officials: DIMITRIOS DRAGANIDIS, PhDc, Principal Investigator — UNIVERSITY OF THESSALY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES
Locations (1):
- Exercise Biochemistry Laboratory, School of Physical Education & Sports Sciences, University of Thessaly, Trikala, Greece